CLINICAL TRIAL: NCT06068894
Title: Safety, Tolerability, and Biosignature of Humanized Prebiotics in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 21-2453
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Intestinal Health
Keywords: Prebiotics; Galactooligosaccharides; Lactosamine

STUDY DESIGN:
Intervention Model Description: 3 arms: GOS, hGOS, or placebo, with 16 participants per arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lactosamine-enriched "humanized" galacto-oligosaccharides (hGOS) (Experimental): The treatment will consist of 10-15 g/day of hGOS, which will be provided to participants as a powder that can be added to any non-alcoholic beverage. The intervention will last for 4 weeks since the research team has shown in adult individuals that a 4-wk period allows for the observation of changes to the gut microbiome. The study will end after the second time-point sample collection at 4 weeks.
  Interventions: Dietary Supplement: "Humanized" galacto-oligosaccharides (hGOS)
- galacto-oligosaccharides (GOS) (Experimental): The treatment will consist of 10-15 g/day of GOS, which will be provided to participants as a powder that can be added to any non-alcoholic beverage. The intervention will last for 4 weeks since the research team has shown in adult individuals that a 4-wk period allows for the observation of changes to the gut microbiome. The study will end after the second time-point sample collection at 4 weeks.
  Interventions: Dietary Supplement: Galacto-oligosaccharides (GOS)
- Placebo (Placebo Comparator): The placebo comparator treatment will consist of 10-15 g/day placebo powder, that can be added to any non-alcoholic beverage. The intervention will last for 4 weeks to mirror the treatment arms. The study will end after the second time-point sample collection at 4 weeks.
  Interventions: Other: Matching Placebo

INTERVENTIONS:
Dietary Supplement: "Humanized" galacto-oligosaccharides (hGOS) — 10-15 g/day of hGOS, which will be provided to participants as a powder that can be added to any non-alcoholic beverage
  Other Names: hGOS
  Arms: lactosamine-enriched "humanized" galacto-oligosaccharides (hGOS)
Dietary Supplement: Galacto-oligosaccharides (GOS) — 10-15 g/day of GOS, which will be provided to participants as a powder that can be added to any non-alcoholic beverage.
  Other Names: GOS
  Arms: galacto-oligosaccharides (GOS)
Other: Matching Placebo — 10-15 g/day powdered corn syrup comprised of fructose, glucose, and an inert cellulose material that matches the consistency, color sweetness, and taste of the prebiotics, that can be added to any non-alcoholic beverage.
  Other Names: Sugar powder
  Arms: Placebo

SUMMARY:
This study aims to establish the safety of a 15 g/day dose of pure prebiotics ß(1-4) galacto-oligosaccharides (GOS) and GOS enriched with N-Acetyl-D-lactosamine, a building block of gut glycoproteins and human milk oligosaccharides (LAcNac, humanized GOS, hGOS) in healthy adult individuals. The safety and tolerability of the dose and the biological signature of GOS and hGOS in healthy adults will be established through a pilot clinical trial to assess GOS and hGOS effects vs placebo on (i) gastrointestinal adverse effects as measured by the Gastrointestinal Symptom and Severity Checklist (GSSC), (ii) increased abundance of beneficial gut bacteria and restoration of the gut microbiome saccharolytic potential, (iii) modulation of biomarkers of inflammation and (iv) evaluation of intestinal barrier function.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be nonsmokers and well-nourished according to standard anthropometric criteria with BMI between 18.5 and 32.
* Individuals must be able to give informed consent.
* Subjects willing and able to:

  * consume prebiotics or placebo preparations for a period of 4 weeks.
  * Record daily food consumption using the Centers for Disease Control and Prevention (CDC) My Food Diary questionnaire.
  * provide stool and blood (via venipuncture) samples.
* Enrollment will not be restricted based on race, ethnicity, or gender. The subject population will reflect the population providing a broad selection of individuals to allow enrollment of subjects from all races, ethnicities, and genders, as represented in North Carolina state.

Exclusion Criteria:

* Less than 18 years of age or older than 55 years of age
* Pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Becker-Dreps, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC-Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty participants signed informed consent and enrolled in the study. Before the baseline visit (Week 0), 10 participants voluntarily withdrew consent, leaving 50 participants who completed the baseline assessment.
Period: Overall Study
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Started | 17 | 17 | 16
Completed | 15 | 15 | 11
Not Completed | 2 | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo | Total
Number analyzed (Participants) | 17 | 17 | 16 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 16 | 50
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 13 | 15 | 13 | 41
  Male | 3 | 2 | 3 | 8
  Non-binary | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 16 | 15 | 14 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 3 | 4 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 12 | 10 | 11 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 17 | 16 | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean Composite PROMIS Maximum Scores
Description: The overall Patient-Reported Outcomes Measurement Information System (PROMIS) score symptom (composite) was calculated as follows: Individual items from the GI questionnaire were grouped into seven symptom domains: abdominal pain, bloating, abdominal distension, flatulence, constipation, diarrhea, and nausea. Each item was rated on a 0-4 scale (0 = "never," 4 = "always"). For each participant at each visit (week 0 and week 4), a domain-specific symptom severity score was defined as the maximum item score within that domain (range 0-4). Using the seven domain severity scores, a composite PROMIS maximum GI measure was calculated for each visit. Composite PROMIS maximum was defined as the maximum severity score cumulatively across all seven domains, representing the participant's worst GI symptoms at that time point. The range of the composite PROMIS maximum score is 0-28 with lower scores representing lowest GI symptoms.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
score on a scale
  Baseline (Week 0) | 4.3 (2.5) | 5.0 (2.3) | 3.0 (2.0)
  Week 4 | 4.4 (1.6) | 3.1 (1.0) | 4.6 (2.1)

2. Secondary Outcome: Mean Percent Change in Relative Abundance of Beneficial Bacteria
Description: The difference in relative abundance of beneficial bacteria of interest include Bifidobacterium and Akkermansia (pre and post intervention) as measured by whole genome sequencing of stool.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
percent change
  Bifidobacterium breve | 0.02 (0.05) | 0.04 (0.09) | -0.01 (0.03)
  Bifidobacterium longum | 1.13 (2.12) | 2.00 (4.05) | -0.23 (0.67)
  Bifidobacterium bifidum | -0.03 (0.16) | 0.51 (1.40) | 0.04 (0.08)
  Bifidobacterium adolescentis | 2.01 (3.91) | 4.96 (7.85) | -0.14 (0.87)
  Bifidobacterium pseudocatenulatum | 1.39 (2.60) | 0.91 (2.37) | -0.42 (1.17)
  Bifidobacterium dentium | 0.01 (0.01) | 0.01 (0.02) | 0.00 (0.00)
  Bifidobacterium catenulatum | 0.24 (0.48) | 0.08 (0.11) | -0.01 (0.04)
  Bifidobacterium pseudolongum | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Akkermansia muciniphila | 0.29 (0.66) | 0.45 (1.78) | -0.23 (0.89)

3. Secondary Outcome: Interleukin-1α Concentration
Description: Modulation of inflammatory biomarker as measured by the MCYTOMAG-70K (Milliplex) reported in pg/mL.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
pg/mL
  Baseline (Week 0) | 1.11 (4.00) | 0.17 (0.52) | 0.00 (0.00)
  Week 4 | 0.40 (0.96) | 0.02 (0.08) | 0.07 (0.16)

4. Secondary Outcome: Interleukin-1ß Concentration
Description: Modulation of inflammatory biomarker as measured by the MCYTOMAG-70K (Milliplex) reported in pg/mL.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
pg/mL
  Baseline (Week 0) | 0.43 (1.25) | 0.15 (0.59) | 0.57 (1.44)
  Week 4 | 0.55 (2.14) | 0.49 (1.30) | 0.33 (1.14)

5. Secondary Outcome: Interleukin-6 Concentration
Description: Modulation of inflammatory biomarker as measured by the MCYTOMAG-70K (Milliplex) reported in pg/mL.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
pg/mL
  Baseline (Week 0) | 1.87 (1.50) | 4.57 (9.70) | 2.56 (1.78)
  Week 4 | 1.87 (1.60) | 3.26 (5.73) | 2.10 (1.82)

6. Secondary Outcome: Interleukin-8 Concentration
Description: Modulation of inflammatory biomarker as measured by the MCYTOMAG-70K (Milliplex) reported in pg/mL.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
pg/mL
  Baseline (Week 0) | 12.86 (6.16) | 11.20 (5.21) | 13.25 (7.19)
  Week 4 | 101.92 (352.85) | 11.53 (5.29) | 14.82 (7.33)

7. Secondary Outcome: Interleukin-12 Concentration
Description: Modulation of inflammatory biomarker as measured by the MCYTOMAG-70K (Milliplex) reported in pg/mL.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
pg/mL
  Baseline (Week 0) | 85.35 (193.49) | 4.60 (11.34) | 14.08 (108.31)
  Week 4 | 9.49 (24.10) | 4.13 (8.10) | 47.19 (100.19)

8. Secondary Outcome: Interleukin-17 Concentration
Description: Modulation of inflammatory biomarker as measured by the MCYTOMAG-70K (Milliplex) reported in pg/mL.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
pg/mL
  Baseline (Week 0) | 17.71 (58.31) | 2.89 (4.81) | 26.96 (80.85)
  Week 4 | 2.88 (6.09) | 6.23 (11.61) | 34.14 (111.18)

9. Secondary Outcome: Interleukin-18 Concentration
Description: Modulation of inflammatory biomarker as measured by the MCYTOMAG-70K (Milliplex) reported in pg/mL.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
pg/mL
  Baseline (Week 0) | 377.68 (114.18) | 464.26 (166.10) | 415.11 (115.77)
  Week 4 | 387.98 (150.25) | 459.46 (140.76) | 412.02 (164.36)

10. Secondary Outcome: Tumor Necrosis Factor Alpha (TNF-α) Concentration
Description: Modulation of inflammatory biomarker as measured by the MCYTOMAG-70K (Milliplex) reported in pg/mL.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
pg/mL
  Baseline (Week 0) | 3.53 (1.48) | 3.98 (2.25) | 4.63 (1.41)
  Wek 4 | 3.68 (1.86) | 4.32 (2.47) | 4.82 (2.17)

11. Secondary Outcome: Interferon Gamma (IFNγ) Concentration
Description: Modulation of inflammatory biomarker as measured by the MCYTOMAG-70K (Milliplex) reported in pg/mL.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
pg/mL
  Baseline (Week 0) | 3.37 (3.27) | 4.04 (3.21) | 5.50 (3.49)
  Week 4 | 3.30 (2.80) | 5.51 (6.75) | 4.05 (2.39)

12. Secondary Outcome: Change in C-Reactive Protein Concentration
Description: Modulation of inflammatory biomarker as measured in serum by commercial enzyme-linked immunosorbent assay (ELISA) kit reported in mg/L.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
mg/L | -0.21 (0.32) | -0.28 (0.35) | -0.03 (0.27)

13. Secondary Outcome: Change in Zonulin Concentration
Description: Used to assess modulation in intestinal barrier function in blood and reported in ng/mL.
Time Frame: Between week 0 (Baseline) and week 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
Number analyzed (Participants) | 15 | 15 | 11
ng/mL | -11.42 (18.45) | 2.15 (21.45) | 6.06 (19.99)

ADVERSE EVENTS:
Time Frame: From Baseline (Week 0) and continued until Week 5, up to a total of 5 weeks.
Arm/Group | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) | Galacto-oligosaccharides (GOS) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 1/17 | 0/17 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactosamine-enriched "Humanized" Galacto-oligosaccharides (hGOS) (N=17) | Galacto-oligosaccharides (GOS) (N=17) | Placebo (N=16)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT06068894/Prot_SAP_000.pdf